CLINICAL TRIAL: NCT01834586
Title: Pilot Study of Anesthetic Topical Adhesive (Synera™) to Reduce Injection Pain With Subcutaneous Multiple Sclerosis Medications (OUCH)
Brief Title: Anesthetic Topical Adhesive (Synera™) to Reduce Injection Pain With Subcutaneous Multiple Sclerosis Medications
Acronym: OUCH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brown, Theodore R., M.D., MPH (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TRB 2012
Record Dates: First submitted 2013-04-02; First posted 2013-04-18 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anesthetic Topical Adhesive Synera (Other): Anesthetic Topical Adhesive Synera. For subjects taking interferon beta subcutaneous (Betaseron, Extavia or Rebif) apply one patch 60 minutes prior to each injection (every-other day or three times per week) for two weeks, then 30 minutes prior for two weeks.
  For subjects taking glatiramer acetate subcutaneous (Copaxone) apply one patch 60 minutes prior to each injection (daily) for one week and then 30 minutes prior for one week.
  Interventions: Drug: Anesthetic Topical Adhesive Synera

INTERVENTIONS:
Drug: Anesthetic Topical Adhesive Synera — For subjects taking interferon beta subcutaneous (Betaseron, Extavia or Rebif) apply one patch 60 minutes prior to each injection (every-other day or three times per week) for two weeks, then 30 minutes prior for two weeks.
  For subjects taking glatiramer acetate subcutaneous (Copaxone) apply one patch 60 minutes prior to each injection (daily) for one week and then 30 minutes prior for one week
  Other Names: Synera

SUMMARY:
The purpose of this study is to see if applying an anesthetic topical adhesive, Synera®, will reduce the injection pain. Relieving injection site pain may improve the tolerability of Multiple Sclerosis medications.

Study Hypothesis: Pre-medication with Synera will have a significant effect on pain ratings as measured by the visual analog scale and Local injection site reaction scale.

DETAILED DESCRIPTION:
Open-label prospective study of Synera to reduce injection pain in 30 patients with relapsing forms of Multiple Sclerosis taking interferon beta or glatiramer acetate. The duration will be 3-6 weeks (1-2 weeks of baseline observation followed by 2-4 weeks of on-drug observation), depending on which Multiple Sclerosis drug product is being studied. The study will include down-titration from 60 to 30 minutes of application to assess for any difference in responses. We define one primary outcome measure,"pain upon injection" by visual analog scale (VAS). Secondary measures will include 24-hour ratings of pain by VAS and 24-hour local injection site reaction (LISR) scale score.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Multiple Sclerosis based on McDonald or Poser criteria (no sub-type restrictions)
* Aged >18
* Regular use of one of the follow Multiple Sclerosis medication treatments: interferon beta subcutaneous (15 subjects, Betaseron, Extavia or Rebif), or glatiramer acetate subcutaneous (15 subjects, Copaxone).
* No change in disease modifying therapy in 60 days.
* Mean score of ≥1.0 on Local Injection Site Reaction scale and Mean Pain Upon Injection score ≥4.0 during baseline period.
* At least 4 valid diary entries over screening period.
* No Multiple Sclerosis exacerbation for 60 days prior to screening.
* Written informed consent

Exclusion Criteria:

* Females who are breast-feeding, pregnant or have potential to become pregnant during the course of the study (fertile and unwilling/unable to use effective contraceptive measures).
* Cognitive deficits that would interfere with the subject's ability to give informed consent or perform study testing.
* Concurrent application of any topical medication to treat injection site reactions from screening through final visit.
* History of allergy to lidocaine, tetracaine or PABA (para-amino benzoic acid) containing products.
* Patients receiving class 1 antiarrhythmic agents (i.e. tocainide, mexiletine)
* Any other serious and/or unstable medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore R Brown, MD, MPH, Principal Investigator — Evergreen Health
Locations (1):
- MS Center at Evergreen Health, Kirkland, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: multiple sclerosis clinic
Groups:
- Anesthetic Topical Adhesive Synera: Anesthetic Topical Adhesive Synera. For subjects taking interferon beta subcutaneous (Betaseron, Extavia or Rebif) apply one patch 60 minutes prior to each injection (every-other day or three times per week) for two weeks, then 30 minutes prior for two weeks.
  For subjects taking glatiramer acetate subcutaneous (Copaxone) apply one patch 60 minutes prior to each injection (daily) for one week and then 30 minutes prior for one week.
  Anesthetic Topical Adhesive Synera: For subjects taking interferon beta subcutaneous (Betaseron, Extavia or Rebif) apply one patch 60 minutes prior to each injection (every-other day or three times per week) for two weeks, then 30 minutes prior for two weeks.
  For subjects taking glatiramer acetate subcutaneous (Copaxone) apply one patch 60 minutes prior to each injection (daily) for one week and then 30 minutes prior for one week
Period: Overall Study
Arm/Group | Anesthetic Topical Adhesive Synera
Started | 30
Completed | 29
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Anesthetic Topical Adhesive Synera
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants] — geographic location
  Participants
    United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Pain Rating
Description: Primary Outcome Measure
  •Change from baseline in rating of pain upon injection, recorded immediately post-injection on a 0-10 Visual Analog Scale (VAS, 10 = worst pain, 0 = no pain)Pain upon injection, recorded immediately post-injection on a 0-10 Visual Analog scale (VAS, 10 = worst pain, 0 = no pain).
Time Frame: baseline and two weeks of treatment
Population: completing participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anesthetic Topical Adhesive Synera
Number analyzed (Participants) | 29
units on a scale | 5.7 (3.2)

2. Secondary Outcome: Average Pain Rating
Description: Average Pain Rating over 24-hours, defined as the average injection-site pain over 24-hours on a 0-10 VAS (0 = no pain, 10 = worst pain).
Time Frame: baseline and two weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Anesthetic Topical Adhesive Synera
Number analyzed (Participants) | 29
units on a scale
  baseline | 2.24 (1.74)
  2 weeks, 30minute application | 1.23 (1.23)
  2 weeks, 60minute application | 1.39 (1.49)

ADVERSE EVENTS:
Arm/Group | Anesthetic Topical Adhesive Synera
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 1/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anesthetic Topical Adhesive Synera (N=30)
dizziness (Nervous system disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes